CLINICAL TRIAL: NCT03721328
Title: A Phase 2 Multicenter Feasibility Trial to Evaluate Safety and Efficacy in Patients Treated for Hip or Knee Prosthetic Joint Infection (PJI) With Alternating Irrigation of Vancomycin Hydrochloride (HCl) and Tobramycin Sulfate in Two-Stage Exchange Arthroplasty
Brief Title: Safety and Efficacy in Patients Treated for Hip or Knee PJI With Vancomycin and Tobramycin Joint Irrigation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osteal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPS-001
Record Dates: First submitted 2018-10-17; First posted 2018-10-26 (Actual); Results first posted 2021-12-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Prosthetic Joint Infection
Keywords: Hip; Knee; Biofilm; Minimum-biofilm-eradication-concentration
MeSH Terms: interventions — Vancomycin; Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental (Experimental): Joint irrigation with vancomycin and tobramycin
  Interventions: Combination Product: vancomycin hydrochloride and tobramycin sulfate

INTERVENTIONS:
Combination Product: vancomycin hydrochloride and tobramycin sulfate — vancomycin hydrochloride and tobramycin sulfate via local irrigation

SUMMARY:
Study Type

Prospective, single-arm, open-label, multicenter (3 to 5 sites), interventional trial.

Primary Study Objective

The objective of the study is to determine the safety profile of local antibiotic irrigation for the treatment of PJI.

Primary Outcome Measure

The overall safety profile is characterized by assessing the incidence of adverse events (AEs), serious adverse events (SAEs), suspected adverse reactions, adverse reactions, and unexpected adverse reactions.

Follow-up

Patients will be assessed for all measures at 3 weeks, 6 weeks, 12 weeks, and 12 months from initial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or greater
* Preoperative diagnosis of PJI of the hip or knee per the 2018 Definition of Periprosthetic Hip and Knee Infection
* Chronic PJI (symptoms lasting at least 4 weeks) per Tsukayama et al.
* Medical clearance for surgery
* Physical and mental ability and willingness to comply with the protocol, including the ability to read and complete required forms, and willingness and ability to adhere to the scheduled follow-up visits and requirements of the protocol

Exclusion Criteria:

* Late acute hematogenous infection per Tsukayama et al.
* Patients for whom a two-stage exchange arthroplasty is not indicated
* Sepsis
* Previously failed single- or two-stage revision arthroplasty for PJI (aseptic revision, polyethylene liner exchange, and/or irrigation and debridement with component retention is allowed)
* Patients with PJI of more than one joint
* Patients on chronic antibiotic therapy (≥ 6 months duration)
* Patients who require therapeutic anticoagulation
* Patients on antiplatelet therapy for whom withholding antiplatelet therapy for any amount of time is contraindicated
* Patients with renal insufficiency/failure (serum creatinine ≥ 2.0 mg/dl)
* Patients with uncontrolled diabetes, defined as: hemoglobin A1C levels > 8.0%
* Patients on immunosuppressive therapy, chemotherapy for malignant disease, or glucocorticoid therapy (e.g. prednisone ≥ 10 mg/day).
* Patients with immunodeficiency (e.g., splenectomy; sickle cell anemia; Stage 3 HIV; primary humoral, bone marrow, or other transplantation.)
* Anticipated or potential patient relocation that may interfere with follow-up examinations
* Allergy to vancomycin HCl or tobramycin sulfate (Note: prior history of Red Man's syndrome is not considered an allergy)
* Patients who are pregnant or planning to become pregnant
* Patients in whom negative pressure wound therapy is contraindicated
* Patients infected with pathogens that are not considered susceptible to vancomycin HCl or tobramycin sulfate, as per the Investigator's opinion
* Breastfeeding at screening visit
* Patients who are prisoners
* Participation in another clinical trial of another Investigational Drug or Investigational Device within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Springer, MD, Principal Investigator — Ortho Carolina Research Institute
Locations (4):
- United States (4):
  - Covenant Hospital, Saginaw, Michigan
  - Ortho Carolina Research Institute, Charlotte, North Carolina
  - SSM Health Bone and Joint Hospital at St. Anthony, Oklahoma City, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Local Irrigation With Vancomycin + Tobramycin: Joint irrigation with vancomycin and tobramycin
  vancomycin hydrochloride and tobramycin sulfate: vancomycin hydrochloride and tobramycin sulfate via local irrigation
Period: Overall Study
Arm/Group | Local Irrigation With Vancomycin + Tobramycin
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.27 (7.329)
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 2
  >= 60 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 14
Region of Enrollment [Number; unit: participants]
  United States | 15
Affected Joint [Count of Participants; unit: Participants]
  Knee | 14
  Hip | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluations: Number and Frequency of Adverse Events Among Participants
Description: The overall safety profile is characterized by assessing the incidence of adverse events (AEs), serious adverse events (SAEs), suspected adverse reactions, adverse reactions, and unexpected adverse reactions.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 15
Participants
  Any Adverse Event | 14
  AE Relationship to NPWT Device UNRELATED | 14
  AE Relationship to Study Medication UNRELATED | 14
  AE Relationship to Study Treatment Procedure UNRELATED | 14
  Severity - Mild | 14
  Severity - Moderate | 7
  Severity - Severe | 6
  Serious Adverse Event | 7
  SAE Relationship to NPWT Device UNRELATED | 7
  SAE Relationship to Study Medication UNRELATED | 7
  SAE Relationship to Study Treatment Procedure UNRELATED | 7
  Suspected Adverse Reaction | 0
  Adverse Reactions | 0

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Local Irrigation With Vancomycin + Tobramycin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Local Irrigation With Vancomycin + Tobramycin (N=15)
Atrial Flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 2
Pulmonary oedema (Cardiac disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Device loosening (Product Issues) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Local Irrigation With Vancomycin + Tobramycin (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1 — General disorders and administration site conditions
Oedema peripheral (General disorders) | 1 — General disorders and administration site conditions
Peripheral swelling (General disorders) | 5 — General disorders and administration site conditions
Pyrexia (General disorders) | 2 — General disorders and administration site conditions
Drug hypersensitivity (Immune system disorders) | 1
Arthritis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Stitch abscess (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 8
Bone contusion (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1
Fungal test positive (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Joint warmth (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Catheter placement (Surgical and medical procedures) | 1
Endodontic procedure (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Wound drainage (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03721328/Prot_SAP_000.pdf